CLINICAL TRIAL: NCT06317038
Title: Performance of TOTAL30 (Lehfilcon A) Contact Lenses in Patients Using Digital Devices and 89814415
Brief Title: To Evaluate the Performance of Total 30 (Lehifilcon A) Contact Lenses in Patients Using Digital Devices for Greater Than 8 Hours Per Day 5 Days Per Week Based on Subjective Reported Data.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tauber Eye Center (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Joseph Tauber, Crystal Remington OD, FAAO, Tauber Eye Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 89814415
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Eye Strain
Keywords: Contact lenses; Digital Devices; Eye Comfort
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Intervention Model Description: Open label Observation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital Device uses for 8 hours per day (Other): Observational responses from patients using digital devices for 8 hours per day will be given a monthly Total 30 Contact lens.
  Interventions: Device: Total 30 Contact Lens

INTERVENTIONS:
Device: Total 30 Contact Lens — Patients will be give a contact lens for 1 month

SUMMARY:
To evaluate the performance of Total 30® (lehfilcon A) contact lenses in patients using digital devices for greater than 8 hours per day 5 days per week based on subjective reported data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-40 of any sex and any race.
* Reports habitually using digital device usage (phone, Ipad, computer, social media, video streaming) for 8 hours or more per day 5 days per week with plans to continue the habit throughout the study.
* Wearing contact lenses for at least 13 hours daily 5 days per week.
* Spherical refractive error between -11.00 D and +6.00D with < -0.75 D of astigmatism.
* Willing to comply with the protocol instructions.
* Has read (or has had read to), understood, and signed an Informed Consent.
* Willing to not use any artificial tears, rewetting drops or dry eye treatments during the study.

Exclusion Criteria:

* Active ocular infection or ocular inflammatory disease.
* Presbyopic or pre-presbyopic that have a measured add power for reading.
* Current Total 30 contact lens wearer.
* Anterior basement membrane dystrophy or history of recurrent erosion syndrome or topographical abnormalities that might indicate ectasia or other corneal degenerative conditions.
* Current or previous diagnosis of dry eye disease; currently using a dry eye treatment including but not limited to artificial tears, rewetting drops or prescription treatments.
* History of severe / serious ocular pathology or other medical conditions that could result in an inability to safely complete the study.
* Participation by the patient in any other investigational study within the past 30 days.
* Unlikely to comply with protocol instructions for any reason (confusion, substance abuse, etc.). The Principal Investigator or the Medical Monitor reserves the right to declare a patient ineligible based on medical evidence that indicates the patient is unsuitable for the study.
* Inability to utilize Clear Care Cleaning solution.
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Likert question about comfort satisfaction while wearing Total 30 contact lenses on a typical day (> 13 hours of daily wear) after 1 month of wear and heavy digital device usage (>8 hours daily wear). | 1 month
  Likert Questionaire: Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree

SECONDARY OUTCOMES:
Likert responses to insertion comfort and overall vision, and heavy digital device use on a typical day after 1 month of wear. | 1 month
  Likert Questionaire: Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree
Results of subjective ratings of patients using Total 30 lenses and heavy digital device usage with VAS diary questionnaire. | 1 month
  VAS diary: scale 0-100 (0=No Discomfort 100= Maximal Comfort)
Report on total daily wear time and digital device usage. | 1 month
  Survey: Total number of hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tauber Eye Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.